CLINICAL TRIAL: NCT05075304
Title: A Phase Ib, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of BDB-001 Injection in Patients With Novel Coronavirus (2019-nCoV) Infection
Brief Title: A Safety and Tolerability Study of BDB-001 in Mild, Moderate COVID-19 Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the COVID-19 epidemic situation, the sponsor has decided to terminate the project.
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Beijing Defengrui Biotechnology Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STS-BDB001-02
Record Dates: First submitted 2021-08-22; First posted 2021-10-12 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BDB001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A low dose of BDB-001 (Experimental): 6 patients administered low dose of BDB-001 injection
  Interventions: Drug: BDB-001 injection
- A intermediate dose of BDB-001 (Experimental): 6 patients administered intermediate dose of BDB-001 injection
  Interventions: Drug: BDB-001 injection
- A high dose of BDB-001 (Experimental): 3-6 patients administered high dose of BDB-001 injection
  Interventions: Drug: BDB-001 injection

INTERVENTIONS:
Drug: BDB-001 injection — IV infusions of Injection diluted in sodium chloride
  Arms: A low dose of BDB-001
Drug: BDB-001 injection — IV infusions of Injection diluted in sodium chloride
  Arms: A intermediate dose of BDB-001
Drug: BDB-001 injection — IV infusions of Injection diluted in sodium chloride
  Arms: A high dose of BDB-001

SUMMARY:
This open, multi-center, multiple ascending dose study was designed to evaluate the safety, tolerability, preliminary efficacy and PK/PD of BDB-001 injection in patients with mild, or general COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ age ≤60, 18 kg/m2 ≤BMI ≤28 kg/m2, male or female;
* Diagnosed with 2019-nCoV infection and classified clinically as mild or general;
* Agreed not to participate in other clinical studies before completing this study;
* With the subject's consent and signed informed consent form by the subject or his/her legal representative.

Exclusion Criteria:

* Diagnosed with 2019-nCoV infection and classified clinically as severe or critical severe; severe pneumonia or acute respiratory distress syndrome, sepsis and septic shock;
* The disease would deteriorate significantly within 48 hours judged by the investigators;
* Immunodeficiency or immune related diseases not suitable for participation judged by the investigators (such as autoimmune diseases, IgG4 related diseases, allergic alveolitis, vasculitis, etc);
* Lymphocyte count <0.5×109/L;
* Neutropenia history (neutrophil absolute count was less than 2×109/L in adults), except for infection;
* D- dimer >2000 µg/L;
* Severe history of lung diseases, such as chronic obstructive pulmonary disease, lung cancer, tuberculosis, etc., history of heart disease: unstable angina pectoris, myocardial infarction, cardiac surgery, cardiac function≥ grade 3 (NYHA classification), serious history of liver disease (such as Child Pugh score ≥grade C), serious renal disease history, such as renal insufficiency (GFR ≤ 15ml/min/1.73m2), etc;
* The subjects used the following drugs within 2 weeks (including 2 weeks) before screening:

  1. Calcineurin inhibitors (such as cyclosporin and tacrolimus);
  2. Proliferation inhibitors (such as everolimus, sirolimus, etc);
  3. anti-metabolic agents (such as mycophenolate mofetil, mycophenolic acid, purine sulfate, etc);
* Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAEs) and non-serious adverse events | Up to Day 40
  An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician. Number of participants who had SAEs and non-SAEs are presented.
Number of participants with abnormal laboratory tests | Up to Day 40
  Blood samples were collected for the assessment of laboratory tests. Number of participants with abnormal laboratory tests parameters are presented.
Number of participants with physical examination | Up to Day 40
  Blood samples were collected for the assessment of physical examination. Number of participants with abnormal physical examination parameters are presented.
Number of participants with abnormal vital signs | Up to Day 40
  Vital signs were measured in a semi-supine position after five minutes of rest and included temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP) , heart rate, respiratory rate. Number of participants with abnormality in any vital signs are presented.
Number of participants with abnormal electrocardiogram (ECG) findings | Up to Day 40
  Number of participants with abnormality Abnormal Electrocardiogram (ECG) are presented.
Plasma concentration of BDB-001 following intravenous administration | Within 60 minutes (prior to start of BDB-001 IV infusion), 10 minutes (end of infusion); at 6, 12,24, 48 hours after end of infusion.
  Blood samples were collected at indicated time points for measurement of Plasma concentrations of BDB-001 following intravenous administration. Pharmacokinetic Population comprised of all participants for whom at least one evaluable pharmacokinetic sample was obtained and analyzed.
Plasma concentration of ADA | Within 60 minutes (prior to start of the first and second BDB-001 IV infusion), Day 7 24 hours after infusion, day 14.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sanya Central Hospital (Hainan Third People'S Hospital), Sanya, Hainan
  - Renmin Hospital Of Wuhan University Bubei General Hospital, Wuhan, Hubei
  - General Hospital of Gentral Rheater Command, Wuhan, Hubei
  - Shu Lan (Hangzhou) Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No